CLINICAL TRIAL: NCT01657006
Title: HeartTrends HRV Algorithm for the Diagnosis of Myocardial Ischemia
Brief Title: HeartTrends Heart Rate Variability (HRV) Algorithm for the Diagnosis of Myocardial Ischemia
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9581-IG-CTIL
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Ischemic Heart Disease
Keywords: Heart rate variability; ischemic heart disease; myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators intend to prospectively enroll consecutive patients, without known ischemic heart disease, referred by their physician for routine exercise MPI at a tertiary care center.

Prior to the MPI (nuclear stress test), eligible and consenting patients will undergo a one-hour period of Holter ECG digital recording. Application of ECG electrodes will be performed by medical technicians following standard recommendations, utilizing approved Holter device & stickers. The Holter ECG data will be used for the offline heart rate variability (HRV) analysis by the HeartTrends device.

Immediately following data acquisition, all patients will undergo an exercise MPI according to accepted clinical practice guidelines.

Following the MPI, there will be no interference with patient management, which will be conducted by the patients' treating physicians according to current guidelines, unaware of HRV results.

Analysis of recorded ECG data for HRV will be performed blinded to the EST and MPI results, by HeartTrends device.

The results of the HRV tests will not be available to treating physicians and will not be used to guide patient management. Patients will be followed for 6 months for the occurrence of coronary interventions and MACE, defined as: death, myocardial infarction, unstable angina, or any coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Referral for exercise MPI by treating physicians
* Willing and able to provide written informed consent

Exclusion Criteria:

* Established ischemic heart disease
* Atrial fibrillation or flutter
* Acute Coronary Syndrome
* Cardiac Pacemaker
* Clinical diagnosis of heart failure
* Moderate or severe COPD
* Active myocarditis, constrictive pericarditis, any cardiomyopathy, cardiac or systemic amyloidosis
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
* Any illness that might reduce life expectancy to less than 1 year from screening
* Left bundle branch block (LBBB), significant intra-ventricular conduction delay (IVCD) or significant (>1mm) ST deviations on baseline ECG
* Inability to perform an exercise stress test (i.e. orthopedical or neurological limitations)
* Any significant established myocardial or valvular disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will prospectively enroll consecutive patients, without known ischemic heart disease, referred by their physician for an exercise MPI.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the HeartTrends device for the detection of myocardial ischemia | 6 month
  sensitivity of the HeartTrends device in comparison to conventional exercise stress testing for the purpose of diagnosing significant myocardial ischemia based on exercise myocardial perfusion imaging examination (considered as the "gold standard")

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Goldenberg I, Goldkorn R, Shlomo N, Einhorn M, Levitan J, Kuperstein R, Klempfner R, Johnson B. Heart Rate Variability for Risk Assessment of Myocardial Ischemia in Patients Without Known Coronary Artery Disease: The HRV-DETECT (Heart Rate Variability for the Detection of Myocardial Ischemia) Study. J Am Heart Assoc. 2019 Dec 17;8(24):e014540. doi: 10.1161/JAHA.119.014540. Epub 2019 Dec 16. PMID 31838969
- [Derived] Goldkorn R, Naimushin A, Shlomo N, Dan A, Oieru D, Moalem I, Rozen E, Gur I, Levitan J, Rosenmann D, Mogilewsky Y, Klempfner R, Goldenberg I. Comparison of the usefulness of heart rate variability versus exercise stress testing for the detection of myocardial ischemia in patients without known coronary artery disease. Am J Cardiol. 2015 Jun 1;115(11):1518-22. doi: 10.1016/j.amjcard.2015.02.054. Epub 2015 Mar 14. PMID 25872904